CLINICAL TRIAL: NCT05444062
Title: Quebec Lung Cancer Screening PLUS Trial - a Randomized Controlled Trial of an Educational Intervention for Untreated Chronic Obstructive Pulmonary Disease (COPD) and/or Cardiovascular Disease (CVD) Identified During Lung Cancer Screening
Brief Title: Quebec Lung Cancer Screening PLUS Trial
Acronym: QLC+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicole Ezer, MD, FRCPC, MPH (Other)
Responsible Party: Sponsor-Investigator, Nicole Ezer, MD, FRCPC, MPH, Assistant professor of medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MP-37-2023-8641
Record Dates: First submitted 2022-06-27; First posted 2022-07-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: COPD; Coronary Artery Calcification
Keywords: COPD; Coronary Artery Calcification; Lung cancer screening; Undiagnosed disease; Educational intervention; Medication adherence; Untreated disease; Statins; Inhalers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Undiagnosed Diseases; Medication Adherence | interventions — General Practitioners; Pharmacists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Arm: CVD (No Intervention): Patients diagnosed with mild to severe CAC and not on first line guideline recommended therapy.
  Coronary artery Calcification (CAC) score obtained from lung cancer screening CT Scan images
- Intervention Arm: CVD (Other): Patients diagnosed with mild to severe CAC and not on first line guideline recommended therapy.
  CAC score obtained from lung cancer screening CT Scan images
  Interventions: Behavioral: Educational material and treatment recommendations for patients, general practitioners and pharmacists
- Control Arm: COPD (No Intervention): Patients with untreated COPD or not on first line guideline recommended therapy.
- Intervention Arm: COPD (Other): Patients with untreated COPD or not on first line guideline recommended therapy.
  Interventions: Behavioral: Educational material and treatment recommendations for patients, general practitioners and pharmacists

INTERVENTIONS:
Behavioral: Educational material and treatment recommendations for patients, general practitioners and pharmacists — Educational material and treatment recommendations given to patients, their family doctors and their pharmacists.
  Arms: Intervention Arm: COPD; Intervention Arm: CVD

SUMMARY:
Does an educational intervention for untreated COPD and cardiovascular disease which is integrated in an existing lung cancer screening program improve guideline concordant medication adherence at 12 months

ELIGIBILITY:
Inclusion Criteria:

* Patient screened for lung cancer as part of the Quebec Lung Cancer Demonstration project by low dose CT scan of the chest.
* Cardiovascular aim: mild to severe CAC identified on low dose CT, not on guideline recommended lipid-lowering therapy.
* COPD aim: diagnosed with COPD, symptomatic (mMRC >=1 or CAT>= 10) and untreated, or not on first line guideline recommended therapy for COPD.

Exclusion Criteria:

* Any participant with a high suspicion of lung cancer, defined as Lung-RADS (Lung Imaging Reporting and Data System) 3 or 4, as this is an inopportune time to initiate new medical therapies.
* Cardiovascular aim: Absent CAC, known clinical atherosclerosis, known former heart surgery, Diabetes Mellitus.
* COPD aim: asymptomatic, or already on appropriate first line COPD therapy.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Guideline concordant statin therapy 1 year following the first low dose CT scan. | 1 year post CT
  Among patients with moderate to severe coronary artery calcifications (CAC) not on a statin at baseline, any statin prescribed for primary prevention at least once in the 1 year following the first low dose CT scan.
  (aim 1)
Guideline concordant inhaler therapy 1 year following the first low dose CT scan | 1 year post CT
  Among patients who have untreated or inappropriately treated COPD at baseline, any long acting muscarinic antagonist inhaler prescribed at least once in the 1 year following the first low dose CT scan (aim 2)

SECONDARY OUTCOMES:
Medication possession ratio (MPR) - Aim 1 | 1 year post CT
  Reflects patient adherence. Days of drug supply over 1 year with cholesterol lowering medication in the previous 1 year from pharmacy dispensation records.
Medication possession ratio (MPR) - Aim 2 | 1 year post CT
  Reflects patient adherence. Days of drug supply over 1 year with guideline concordant inhaler therapy for COPD in the previous 1 year from pharmacy dispensation records.
COPD Symptoms | Baseline, 6 months post intervention, 12 months post intervention
  COPD Assessment Test is a validated patient-reported outcome. It measures 8 symptoms of COPD on a 0-5 point scale at baseline, 6 and 12 months post intervention
Quality of life using SF-36 questionnaire | Baseline, 12 months post intervention
  SF-36 questionnaire will be filled at baseline and 12 months post intervention
Patient satisfaction with communication and decision making | 3 months post intervention
  COMRADE is a 20-item self-reported measure for use in primary care to assess risk communication and confidence in treatment decision making. It assesses patient satisfaction with information provided about risks/benefits of treatment, perception of participation in treatment decisions, and satisfaction with that decision.
  COMRADE questionnaire will be sent to patients after their first meeting with their general practitioner up to 3 months after intervention.
Health Care Utilisation | 1 year post intervention
  Number of unplanned clinic visits, hospitalizations for respiratory or cardiac disease, consultations with specialists (cardiology and respirology), invasive/non-invasive cardiac or respiratory investigations
Absenteeism and presenteeism | baseline
  Work productivity and activity impairment (WPAI) questionnaire
Health literacy | baseline
  Health literacy will be assessed at study entry using the Brief Health Literacy Screen.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No